CLINICAL TRIAL: NCT06942819
Title: Magnetic Resonance Imaging (MRI) Outcomes of VersaWrap Verve Protector Following Lumbar Decompression Surgery
Brief Title: MRI Outcomes of VersaWrap Nerve Protector Following Surgery
Status: Enrolling by invitation | Type: Observational
Sponsor: Research Source (Network)
Responsible Party: Sponsor
Other Study IDs: TP-081
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Lumbar Decompression
Keywords: VersaWrap; Decompression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- VersaWrap: All enrolled patients will receive VersaWrap Nerve Protector prior to surgical closure
  Interventions: Device: VersaWrap Nerve Protector

INTERVENTIONS:
Device: VersaWrap Nerve Protector — VersaWrap Nerve Protector is applied to the nerve root to protect the surrounding tissues

SUMMARY:
The purpose of this study is to evaluate enhancement patterns in magnetic resonance imaging (MRI) evidence following the use of VersaWrap in bilateral lumbar decompression surgeries.

DETAILED DESCRIPTION:
This study is a prospective, post-market, observational multi-center evaluation of the use of VersaWrap. Patients identified by the Investigator in their practice as needing a bilateral lumbar decompression at one level (L4-S1) and meeting all the inclusion and none of the exclusion criteria. Patients will consent to participating in the study, prior to any study procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 and ≤65 at time of surgery
2. Patients undergoing lumbar decompression bilaterally at one level from L4-S1
3. Psychologically, mentally and physically able to fully comply with this protocol including adhering to follow-up schedule, study requirements with a signed informed consent.

Exclusion Criteria:

1. Non-English speaking
2. Known allergy or sensitivity to citrate, alginate or hyaluronate
3. Known allergy or sensitivity to MRI contrast dye
4. Known to experience claustrophobia
5. Pregnant or breastfeeding at time of surgery
6. Incarcerated at time of surgery
7. Prior lumbar surgery at the index level
8. Conjunction device use at index level (i.e., Barricade)*
9. Patient has any condition, that in the opinion of the Investigator, would prohibit the patient from complying with the protocol *Note: conjunction medications (i.e., Depo-Medrol, Marcaine/Epinephrine) are acceptable

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who meet the following criteria and none of the exclusion will be enrolled in the study. A patient is considered enrolled upon successful placement of VersaWrap during the surgical procedure. If the surgeon decides intra-operatively not to utilize VersaWrap then the patient will be considered a screen failure.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
MRI | 4 months
  Magnetic resonance imaging (MRI) will be used to evaluate enhancement patterns

CONTACTS AND LOCATIONS:
Locations (1):
- Austin Neurosurgeons, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No